CLINICAL TRIAL: NCT04558242
Title: Evaluation of the GENIX, a Low Level Light Device as a Primary Therapy for Androgenetic Alopecia in Men and Women
Brief Title: Low Level Light Device as a Primary Therapy for Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kiierr International, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUAL6594
Record Dates: First submitted 2020-09-14; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Androgenetic Alopecia; Hair Loss; Thinning Hair; Balding
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Genix LLLT Therapeutic Cap (Active Comparator): This is a low-level light device containing 150, 650 nanometer LEDs and 50, 940 nanometer LEDs of equal energy output, fixed at 10 milliwatts in a low profile helmet.
  Interventions: Device: Genix
- Sham Non-therapeutic Placebo Cap (Sham Comparator): Sham Placebo Cap low profile helmet containing no low-level light.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Genix — Low Level Light (LEDs)
  Arms: Genix LLLT Therapeutic Cap
Device: Sham — Incandescent Bulbs Colored Red
  Arms: Sham Non-therapeutic Placebo Cap

SUMMARY:
The purpose of this research is to study the safety and effectiveness of a light therapy device for human hair growth. This device, called the GENIX, is a type of cold, or non-heat producing light emitting diode (LED) that will emit light on the hair growth cells within and around the hair follicle. When these cells do not function properly, one may experience common problems such as baldness and thinning or brittle hair. The application of a special category of low-level non-laser light to be studied in the project may cause an increase in essential nutrients to the damaged hair follicles and skin cells, leading to a reduction in hair loss and in some cases, possibly leading to re-growth.

DETAILED DESCRIPTION:
The application of low-level light therapy has aroused considerable research interest in recent years for the treatment of a variety of clinical indications. These range from pain management to wound healing and most recently to hair regrowth. All have demonstrated biological effects in living organisms. In 1967 Endre Mester, a physician practicing in Budapest Hungary, decided to test the effects of laser radiation on mice and its possible link to resultant cancer. To his great surprise, the mice regrew the shaved hair in half the time of non-radiated mice. This was the first reference to LLLT and hair growth.

This study on LLLT, aims to confirm the established safety and physiologic effects that occur when the human hair follicle and surrounding tissue structures are exposed to this type of radiation. Thus far, all reports on the efficacy of low level light therapy (LED) in this area, have been, in large part, consistent in outcome results, as supported by multi-center, randomized, double blind, controlled studies. This has been in the form of analysis of the non-radiated and radiated tissues as determined by terminal hair counts from baseline to post treatment counts. The theory that is widely accepted is that the mitochondria are the powerhouse of the stem cells that cause hair growth. The LLLT "turns on" the nutrient pump process that energizes the mitochondria, which leads to an increase in ATP and subsequent reversal of hair follicles from the dormant stage of growth called telogen, to the active growth stage called anagen.

This specific light system is unclassified by the FDA, from a radiation standpoint, because the agency has not developed class designations for LEDs. Currently, it is classified as a class II medical device and will be designated as an Over-the-Counter device. It may be marketed for hair regrowth, as defined by an increase in terminal hairs and wellness, which can be defined as thicker, denser, more supple and darker hair shafts.

ELIGIBILITY:
Inclusion Criteria:

* Males- age 18-50, females 18 - 70 having Fitzpatrick skin types I-VI.
* Androgenetic alopecia by history and clinical examination. Norwood-Hamilton Class (IIa-V) and Ludwig-Savin I-II
* Having good health and not belonging to any risk group for possible immunodeficiency of other chronic systemic diseases that affect hair.
* Have a healthy scalp with no anatomical abnormality or suffering with any cutaneous disorder that would preclude participation in this study. Subjects suffering with dermatological conditions such as seborrheic dermatitis or psoriasis can participate provided the scalp is not involved, and no topical treatment is being administered to the scalp during the expected period of treatment.
* Willingness to answer questions related to Safety and Adverse Effects after each treatment.
* Willingness to have the required physical examination performed, for the purpose of evaluating general health.
* Willing to refrain from using any other topical preparation to restore hair, or be involved in any treatment aimed at hair restoration. Having participated in any such treatment will require a 4-week washout period before commencing study.

Exclusion Criteria:

* Family history of malignant melanoma, or any cutaneous cancer in the head and neck area.
* Past medical history of malignant melanoma, or other cutaneous neoplasm in the head and neck area.
* Past Medical History or Family History of Alopecia Areata, or other causes of alopecia, or cancer.
* Past medical history of collagen-vascular disease, thyroid disease or other cutaneous or systemic disease that seriously affects the scalp. (Seborrheic dermatitis or psoriasis under good control with therapy and without showing scalp involvement and not requiring topical scalp therapy would not be a contraindication.)
* Severe androgenetic alopecia (beyond Norwood-Hamilton V or Ludwig-Savin II).
* Previous scalp surgery or signs of any scar on the scalp.
* Taking chemotherapeutic agents, bronchodilators, decongestants, antiepileptic, systemic steroids, topical steroids on the scalp or on greater than 10% body surface area or any medication known to cause hair growth.
* Having any chronic eye illness, including cataracts, glaucoma, any form of retinal eye disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Terminal Hair Growth | 24 Weeks
  Terminal hairs from pre-treatment photographs and post-treatment photographs, as defined by the universally accepted description of a terminal hair shaft of the human scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bodian, MD, Principal Investigator — Bodian Dermatology Group
Locations (1):
- NST Consultants, Inc., Mendham, New Jersey, United States